CLINICAL TRIAL: NCT04896177
Title: A Prospective, Multicenter, Randomized Controlled, Non-inferior Clinical Trial to Evaluate the Efficacy and Safety of Sirolimus Drug-eluting Coronary Balloon Catheter in Treatment of Coronary Bifurcation Lesions
Brief Title: Sirolimus DEB in Coronary Bifurcation Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SalubrisDEB001
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Coronary Bifurcation Lesions
Keywords: drug-eluting balloon; coronary bifurcation lesions; coronary heart disease; sirolimus
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus drug-eluting coronary balloon catheter (Experimental): Manufacturer: Shenzhen Salubris Pharmaceuticals Co., Ltd. This product is a sirolimus drug eluting balloon catheter for coronary artery therapy. It is a rapidly exchangeable PTCA balloon catheter (RX), effective length is 140cm, and compatible with 0.014 in. (0.36mm) guide wire. The balloon at the distal end of the catheter was coated with sirolimus, an anti-proliferative and anti-inflammatory drug.
  Interventions: Device: Sirolimus drug-eluting coronary balloon catheter
- Drug-eluting balloon catheter (Active Comparator): Manufacturer: Liaoning Yinyi Biotechnology Co., Ltd Coated with paclitaxel.
  Interventions: Device: Paclitaxel drug-eluting coronary balloon catheter

INTERVENTIONS:
Device: Sirolimus drug-eluting coronary balloon catheter — Patients in experimental group will undergo PCI, using sirolimus drug-eluting coronary balloon catheter.Subjects without stent implantation were regularly treated with dual antiplatelet for 9 months after surgery. Subjects with stents were regularly treated with dual antiplatelet for 12 months after the surgery, in accordance with the applicable guidelines for percutaneous coronary intervention.
  Arms: Sirolimus drug-eluting coronary balloon catheter
Device: Paclitaxel drug-eluting coronary balloon catheter — Patients in control group will undergo PCI, using paclitaxel drug-eluting coronary balloon catheter.Subjects without stent implantation were regularly treated with dual antiplatelet for 9 months after surgery. Subjects with stents were regularly treated with dual antiplatelet for 12 months after the surgery, in accordance with the applicable guidelines for percutaneous coronary intervention.
  Arms: Drug-eluting balloon catheter

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sirolimus drug-eluting coronary balloon catheter in treatment of coronary bifurcation lesions.

This is a prospective, multicenter, randomized controlled, non-inferior clinical trial, which would enroll 280 participants in total. Paticipants would undergoing PCI with sirolimus DEB or paclitaxel DEB, and be followed-up to 24 months.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of sirolimus drug-eluting coronary balloon catheter in treatment of coronary bifurcation lesions.

This is a prospective, multicenter, randomized controlled, non-inferior clinical trial, which would enroll 280 participants in total. Paticipants with would undergoing PCI with sirolimus DEB or paclitaxel DEB, and be followed-up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female that ages 18-85 year old;
2. Having evidence of myocardial ischemia;
3. Voluntarily participates in this study and signs the informed consent form (ICF);
4. Sufficiently compliant with the study protocol and agreed to receive follow-up at 1 month ±7 days, 6 months ±14 days, 9 months ±30 days, 12 months ±30 days, and 24 months ±30 days, of which angiography was required at 9 months ±30 days;
5. Angiography confirmed as de novo bifurcation lesion with side-branch stenosis (diameter) ≥70%;
6. Suitable for PCI and side-branch lesions are not expected to stent implantation, and no drug-eluting balloon used for the main-branch. If a stent is implanted into the main-branch, it's usually necessary to perform a final balloon kissing on the two branches;
7. Residual stenosis of the side-branch lesion ≦50% after pre-treatment, with a TIMI flow grade 3;
8. The target vessel diameter was 2.0mm-4.0mm.

Exclusion Criteria:

1. Women who is pregnant or lactating, or having a fertility plan within 1 year or are unwilling to take effective contraceptive measures;
2. Cardiogenic shock patients;
3. With hemorrhagic symptoms or active gastrointestinal ulcers, or previous stroke within 6 months, or who are expected to be unable to tolerate double-antibody therapy after interventional therapy;
4. ST-segment elevation myocardial infarction (STEMI) occurred within one week before enrollment;
5. With severe congestive heart failure or NYHA class Ⅳ heart failure;
6. With severe valvuar heart disease;
7. Heart transplant patients;
8. With renal insufficiency (creatinine > 3.0mg/ dL or 265.2 umol /L) and/or advanced renal disease requiring dialysis;
9. With a life expectancy less than 1 year;
10. With contraindications who cannot take aspirin and/or clopidogrel and/or ticagrelor;
11. With known allergies to paclitaxel, sirolimus, contrast agents, etc.;
12. Participating in clinical trials of other drugs or devices and has not met the primary endpoint;
13. Non-target lesions cannot be processed before the target lesions or non-target lesions treatment fails;
14. Intra-stent restenosis;
15. High-risk left main disease;
16. Other patients considered by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
Stenosis of lumen diameter of target lesion branch | 9 months (±30 days)
  The degree of lumen diameter stenosis (%) =(1- the minimum lumen diameter of the vessel/the reference diameter of the target lesion vessel)×100%

SECONDARY OUTCOMES:
Success rate of interventional treatment | Index Procedure
  Including device success, pathological success and clinical success
Incidence of restenosis of target lesions | 9 months (±30 days)
  Restenosis defined as angiographic stenosis ≥50%
Late lumen loss (LLL) | 9 months (±30 days)
Target lesions revascularization (TLR) | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), 24 months (±30 days)
  Including PCI re-stenting, balloon dilation, plaque grinding or excision, coronary artery bypass grafting (CABG)
Target vessel revascularization (TVR) | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), 24 months (±30 days)
  Including PCI re-stenting, balloon dilation, plaque grinding or excision, coronary artery bypass grafting (CABG)
Target lesion failure rate (TLF) | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), 24 months (±30 days)
  Including cardiac death, target vascular-associated myocardial infarction, and target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided